CLINICAL TRIAL: NCT04586088
Title: Apatinib Combined With Camrelizumab in Recurrent or Metastatic Nasopharyngeal Carcinoma Who Failed at Least the First-line Treatment
Brief Title: Apatinib and Camrelizumab in Recurrent or Metastatic Nasopharyngeal Carcinoma With First-line Treatment Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Proffessor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2020-2103
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent Nasopharyngeal Carcinoma; Metastatic Nasopharyngeal Carcinoma; Chemotherapy Effect; Immunotherapy; Molecular Targeted Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus Camrelizumab arm (Experimental): Subjects receive apatinib plus camrelizumab
  Interventions: Drug: Apatinib plus Camrelizumab

INTERVENTIONS:
Drug: Apatinib plus Camrelizumab — Subjects receive Apatinib, 250mg, QD and Camrelizumab, 200mg, D1, Q3W. Treatment was continued until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, or investigator decision.

SUMMARY:
This is a prospective phase II clinical trial to evaluate the efficacy and safety of apatinib and camrelizumab in recurrent or metastatic nasopharyngeal carcinoma who failed at least the first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-70 years of age.
2. Subjects diagnosed with pathological confirmed metastatic nasopharyngeal carcinoma, or subjects with recurrent NPC that is unfit for local treatment
3. Underwent at least first-line treatment failure
4. ECOG performance status of 0 or 1.
5. Life expectancy more than 12 weeks.
6. Subjects enrolled must have measurable lesion(s) according to response evaluation criteria in solid (RECIST) v1.1.
7. Adequate organ function assessed by laboratory parameters during the screening period.
8. Female subjects agree not to be pregnant or lactating from beginning of the study screening through at least 3 months after receiving the last dose of study treatment. Both men and women of reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy.
9. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval;
2. Known history of hypersensitivity to any components of the Camrelizumab formulation or other monoclonal antibodies ;
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses 10 mg/day prednisone or equivalent are prohibited within 4 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed;
4. Subjects who underwent anti-PD-1 /PD-L antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell synergistic stimulation or checkpoint pathway) and anti-angiogenic drugs.
5. Abnormal coagulation function (INR>1.5×ULN, APTT>1.5×ULN) with bleeding tendency.
6. The laboratory test values within 7 days before enrollment do not meet the relevant standards.
7. Active central nervous system (CNS) metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease);
8. Diagnosed with other malignant tumors.
9. Uncontrolled clinically significant medical condition, including but not limited to the following:

   1. Hypertension that cannot be reduced to the normal range after antihypertensive drug
   2. congestive heart failure (New York Health Authority Class > 2),
   3. unstable angina,
   4. myocardial infarction within the past 12 months,
   5. clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
10. Active bleeding, ulcer, intestinal perforation, major surgery in the previous month; Patients with tumors close to the internal carotid artery or other large vessels, thus at risk of massive bleeding
11. Active infection or an unexplained fever; 38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled);
12. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease; active tuberculosis (TB), anti-TB treatment is ongoing or within 1 year prior to screening; Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-Hepatitis B core antibody.
13. Received any anti-infective vaccine (e.g. influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment.
14. Any other medical (eg, pulmonary, metabolic, congenital, endocrinal, or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  Defined as the proportion of patients whose tumors shrink to complete response (CR) or partial response (PR) and remain for a certain period of time according to RECIST 1.1

SECONDARY OUTCOMES:
The proportion of patients who achieved disease control | 1 year
  Defined as the proportion of subjects who achieve CR+PR+stable disease (SD) for at least 4 weeks according to RECIST 1.1.
The proportion of patients who achieved clinical benefit | 1 year
  Defined as maintaining the efficacy of CR+PR+SD for at least 6 months according to RECIST 1.1.
median progression-free survival | 1 year
  Defined as the period from the start of enrollment until disease progression or death from any cause.
Duration of response | 1 year
  Defined as the time from the first assessment of CR and PR to the first assessment of PD or death caused by any cause according to RECIST 1.1.
Adverse events | 1 year
  NCI-CTC5.0 standard was adopted, and the safety was assessed mainly by clinical laboratory tests, ECOG-PS score, physical examination, electrocardiogram, and adverse event results.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ding X, Zhang WJ, You R, Zou X, Wang ZQ, Ouyang YF, Peng L, Liu YP, Duan CY, Yang Q, Lin C, Xie YL, Chen SY, Liu YL, Gu CM, Xie RQ, Huang PY, Hong MH, Hua YJ, Chen MY. Camrelizumab Plus Apatinib in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma: An Open-Label, Single-Arm, Phase II Study. J Clin Oncol. 2023 May 10;41(14):2571-2582. doi: 10.1200/JCO.22.01450. Epub 2023 Feb 3. PMID 36735896